CLINICAL TRIAL: NCT03537222
Title: Validation of the Myeloma Patient Outcome Scale (MyPOS) Assessing the Quality of Life in Patients With Multiple Myeloma in the German Speaking Part of Switzerland
Brief Title: Quality of Life in Patients With Multiple Myeloma-validation Study
Status: Terminated | Type: Observational
Why Stopped: Not enough participants and study funding
Sponsor: Zurich University of Applied Sciences (Other)
Collaborators: Kantonsspital Münsterlingen (Other); Kantonsspital Aarau (Other); Klinik Hirslanden, Zurich (Other); Celgene Corporation (Industry); King's College London (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Julia Dratva, Head of health sciences research unit, Zurich University of Applied Sciences
Other Study IDs: 97107155001701
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Multiple Myeloma
Keywords: quality of life; psychometrics
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MyPOS
  Interventions: Diagnostic Test: Myeloma Patient Outcome Scale (MyPOS)

INTERVENTIONS:
Diagnostic Test: Myeloma Patient Outcome Scale (MyPOS) — Patients complete the MyPOS questionnaire on quality of life

SUMMARY:
In this study, the Myeloma Patient Outcome Scale (MyPOS) will be translated from English to German. This translated version will be quantitatively and qualitatively validated with patients with multiple myeloma.

DETAILED DESCRIPTION:
Patients with multiple myeloma (N=10) will be interviewed in the qualitative phase about their comprehension of the translated MyPOS. The questionnaire will be revised according to the results of the interviews. This culturally adapted Swiss-German MyPOS will be assessed in the quantitative phase for its' psychometric properties with 200 patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* informed consent as documented by signature
* confirmed histological diagnosis of multiple myeloma,
* age ≥ 18 years,
* mental capacity to give written informed consent

Exclusion Criteria:

* inability to communicate in German
* participation in another clinical study
* more than one cancer diagnosis
* mental illness (i.e. psychiatric diagnosis)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Psychometric properties of the culturally-adapted Swiss-German Myeloma Patient Outcome Scale (MyPOS) | upon enrollment
  The primary outcome will be the scores on each item of the culturally-adapted Swiss-German MyPOS. Items are scored on a five-point Likert scale. For the analysis, the three subscales "Symptoms" (range: 0-52), "Emotions" (range:0-68) and "Healthcare Support" (range: 0-12) are assessed as well as the MyPOS total score (range: 0-132 ) by summing up the item scores ranging from 0-4. Higher scores reflect worse quality of life.
  The scores will be used to evaluate the psychometric properties of the culturally-adapted Swiss-German MyPOS:
  * Structural validity,
  * Internal consistency,
  * Construct validity,
  * Convergent and divergent validity.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Dratva, Prof.Dr.med, Principal Investigator — Zurich University of Applied Sciences
Locations (3):
- Switzerland (3):
  - Kantonsspital Aarau, Aarau, Canton of Zurich
  - Kantonsspital Münsterlingen, Münsterlingen, Thurgau
  - Onkozentrum Hirslanden, Zurich